CLINICAL TRIAL: NCT05273944
Title: A Randomized, Open-label, Single-dose, Two-preparation, Two-sequence, Two-cycle Crossover, Bioequivalence Study of Doxorubicin Hydrochloride Liposome Injection in Patients With Breast Cancer/Ovarian Cancer
Brief Title: Bioequivalence Study of Doxorubicin Hydrochloride Liposome Injection (Lipodox®) in Chinese Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Kangzhe Pharmaceutical Co., Ltd. (Industry)
Collaborators: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Hunan Cancer Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); First Affiliated Hospital of Jinan University (Other); Zhejiang Provincial People's Hospital (Other); Yuncheng Central Hospital (Other); Shantou Central Hospital (Other); Yuebei People's Hospital (Other); Cancer Hospital of Guizhou Province (Other); Guangzhou Panyu Central Hospital (Other); Dongguan People's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DHLI-BC/OC-BE-001
Record Dates: First submitted 2022-02-10; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference product-R (Active Comparator): Caelyx® (Janssen-Cilag International NV); 20 mg/10 mL (50 mg/m2 dose). As this is a crossover study, subjects receiving the Reference Product (Caelyx®) in Cycle 1, will receive the Test Product (Lipodox®) in Cycle 2. Cycle is defined as 28-42 days (RT).
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection
- Test Product-T (Experimental): Lipodox® (Sun Pharmaceutical Industries Ltd.); 20 mg/10 mL (50 mg/m2 dose). As this is a crossover study, subjects receiving the Test Product (Lipodox®) in Cycle 1, will receive the Reference Product (Caelyx®) in Cycle 2. Cycle is defined as 28-42 days (TR).
  Interventions: Drug: Doxorubicin Hydrochloride Liposome Injection

INTERVENTIONS:
Drug: Doxorubicin Hydrochloride Liposome Injection — 50mg/m2, intravenous drip on Day 1 of each cycle. On Day 1 of Cycle 1 patients will receive either reference or test product. On Day 1 of Cycle 2, patients will crossover to the alternate reference or test formulation. To measure pharmacokinetic paratemers of Caelyx® versus Lipodox®.
  Other Names: Caelyx®/Lipodox®

SUMMARY:
Bioequivalence study is proposed to be carried out on patients of breast cancer/ ovarian cancer, who are administrated for Doxorubicin Hydrochloride Liposomal Injection Lipodox® or Caelyx® in a dose of 50 mg/m2.

DETAILED DESCRIPTION:
This study is a randomized, open-label, single-dose, two-preparation, two-sequence, two-cycle crossover bioequivalence study. This study will be conducted in female subjects aged 18 to 75 years diagnosed with breast cancer/ ovarian cancer. Each subject will be randomized to two treatment sequences (RT or TR) with equal numbers of patients according to a randomization scheme prepared to start of the trial. The cleaning period was 28-42 days. Serial blood samples for determination of free and liposomal encapsulated doxorubicin plasma concentration for PK analysis will be obtained in each cycle. Blood samples to be obtained at 0 h (within 60 min) before infusion, 15 min, 30 min, 45 min, 60 min, 75 min, 90min after the beginning of infusion, 15 min, 30 min, 1.0 h, 3.0 h, 5.0 h, 8.0 h, 16.0 h, 24.0 h, 36.0 h, 48.0 h, 96.0 h, 168.0 h, 240.0 h, 336.0 h after infusion completed.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects fully understand the purpose, nature, methods and possible adverse reactions of the study, voluntarily participate in the study, and sign informed consent before the study procedure begins;
2. Adult female subjects between 18 to 75 years of age (both inclusive) at the time of screening visit. Body weight is greater than or equal to 40.0 kg. Body surface area (BSA) is less than 1.8 m2;
3. Subjects with histologically or cytological proven: 1) Advanced ovarian cancer patients who had previously failed first-line platinum-containing chemotherapy; Or 2) metastatic breast cancer;
4. ECOG performance status ≤ 2;
5. Life expectancy of at least 3 months;
6. Adequate renal, hepatic function:

   1. Neutrophils ≥1.5×109/L;
   2. Leukocyte≥3×109/L;
   3. Platelet count ≥ 80×109/L;
   4. Hemoglobin (Hb) ≥ 90g/L;
   5. Serum creatinine ≤ 1.5 x ULN;
   6. AST ≤ 2.5 x ULN, ALT ≤ 2.5 x ULN (for liver metastasis≤ 5 x ULN);
   7. Prothrombin time (PT)/activated partial thromboplastin time (APTT) ≤ 1.5 x ULN;
   8. Total bilirubin≤ 1.5 x ULN (for liver metastasis≤ 3 x ULN);
   9. Alkaline phosphatase ≤ 2.5 x ULN;
7. Subjects (including spouse) who have no childbearing plans in the next 6 months and voluntarily take effective contraceptive measures.

Exclusion Criteria:

1. History of allergy to doxorubicin or any components of doxorubicin; or those with allergic constitution: such as those who are allergic to two or more drugs and food;
2. Previous treatment with Doxorubicin Liposome, and discontinue treatment due to treatment failure or severe adverse reactions;
3. Patients who have previously received more than 400 mg/m2 doxorubicin (Conversion of other anthracyclines and anthraquinone: 1 mg doxorubicin is equivalent to 2 mg epirubicin, or 2 mg pirarubicin, or 2 mg daunorubicin, or 0.5 mg dimethoxy-daunorubicin , or 0.45 mg mitoxantrone), or severe cardiotoxicity from prior exposure to anthracyclines;
4. Positive history of known spinal cord compression or brain metastases (unless asymptomatic, stable for more than 4 weeks, steroid treatment was discontinued at least 4 weeks prior to first administration of Lipodox®/ Caelyx®, and no radiographic evidence of significant edema around the tumor lesion). Untreated patients with disease progression due to brain metastases in the last treatment prior to screening;
5. Subjects with other known active malignancies that require treatment within 5 years;
6. Patients with abnormal cardiac function: ECG examination, QTc>480ms; left ventricular ejection fraction(LVEF)<55%；congestive heart failure, myocardial infraction, or uncontrolled angina pectoris of New York Heart Society≥2 within 6 months prior to enrollment; have undergone heart bypass surgery; Tropoin≥1.5 x ULN；N-terminal brain natriuretic peptide ≥1.5 x ULN; The investigator evaluated the overall cardiac function of the subjects by integrating all examination items.
7. Patients with poor control of hypertension (systolic≥160 mmHg, diastolic>80 mmHg;
8. Diabetes blood glucose control is not up to standard, fasting blood glucose >11.1 mol/L, or accompanied by diabetic complications (diabetic nephropathy, peripheral neuropathy);
9. Radiation therapy or chemotherapy drugs (paclitaxel, cyclosporine, dexrazoxane, cytarabine, streptozotocin, etc.) within 4 weeks before study administration prior to administration, or other anti-tumor therapies such as endocrine therapy, traditional Chinese medicine, and local radiation therapy to relieve pain;
10. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug, or plan to undergo major surgery during the study period and those who have undergone surgery that may affect drug absorption, distribution, metabolism, and excretion;
11. Use of drugs that induce or inhibit liver drug enzymes in the previous 4 weeks prior to administration and during the study (such as: Barbiturates, carbamazepine, phenytoin, griseofulvin);
12. The special diet within 7 days before the study administration may affect drug absorption, distribution, metabolism and excretion during the study, including but no limited to: taking special diets that may image drug metabolism including dragon fruit, mango, grapefruit, lime, carambola, chocolate, or by the preparation of food or drink, or a diet containing caffeine, xanthine, etc;
13. Patients who consumed excessive amounts of tea, coffee, and/or caffeine-rich beverages (more than 8 cups, one cup=250mL) daily for 3 months prior to administration;
14. Patients who smoked more than 5 cigarettes per day during the 3 months prior to administration, or who did not agree to refrain from using any tobacco products during the study;
15. Drinking more than 14 units of alcohol per week in the 3 months prior to administration (1 unit of alcohol≈360mL beer or 45mL 40% alcoholic spirits or 150mL wine);
16. Pregnant women, breast-feeding women or women of childbearing age who are screened for positive pregnancy tests, or who do not agree to use effective contraceptive measures during the trial or whose spouse plans to give birth within 6 months;
17. Patients with positive hepatitis B virus surface antigen (HBsAg) test results and HBV-DNA ≥104 copy number or ≥2000IU/ML, or those with other active infectious diseases (such as hepatitis C, syphilis, or human immunodeficiency virus HIV infection);
18. Subjects who received vaccine within 1 month prior to administration;
19. Previous history of drug abuse;
20. Patients who cannot withstand venipuncture, have a history of needle sickness and blood sickness, or have difficulty in venous blood collection;
21. Patients who had donated blood or lost blood of ≥400mL within 3 months prior to administration, or intended to donate blood (including blood components) during 3 months after the study;
22. The investigator determined that subjects were unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Cmax | Pre-dose (within 60 minutes), 15,30, 45,60,75,90minutes after the beginning of infusion, 15minutes, 30minutes, 1,3,5,8,16,24,36,48,96,168,240,336hours after infusion completed
  Maximum observed plasma concentration
AUC[0-t] | Pre-dose (within 60 minutes), 15,30, 45,60,75,90minutes after the beginning of infusion, 15minutes, 30minutes, 1,3,5,8,16,24,36,48,96,168,240,336hours after infusion completed
  Area under the plasma concentration-time curve from time 0 to last time of quantifiable concentration
AUC[0-∞] | Pre-dose (within 60 minutes), 15,30, 45,60,75,90minutes after the beginning of infusion, 15minutes, 30minutes, 1,3,5,8,16,24,36,48,96,168,240,336hours after infusion completed
  Area under the plasma concentration-time curve from 0 extrapolated to infinite time

SECONDARY OUTCOMES:
AUC[0-48hours] | Pre-dose (within 60 minutes) , 15, 30, 45, 60, 75, 90minutes after the beginning of infusion, 15 minutes, 30 minutes, 1, 3, 5, 8, 16, 24, 36, 48hours after infusion completed
  Area under the plasma concentration-time curve from time of intake until 48hours post-dose
AUC[48hours-t] | 48hours post-dose to the 336hours post-dose
  Area under the plasma concentration-time curve from time of 48hours post-dose until the 336hours posy-dose
Tmax | Pre-dose (within 60 minutes), 15,30, 45,60,75,90minutes after the beginning of infusion, 15minutes, 30minutes, 1,3,5,8,16,24,36,48,96,168,240,336hours after infusion completed
  Time to reach the maximum observed plasma concentration
λz | Pre-dose (within 60 minutes), 15,30, 45,60,75,90minutes after the beginning of infusion, 15minutes, 30minutes, 1,3,5,8,16,24,36,48,96,168,240,336hours after infusion completed
  Elimination rate constant
t1/2z | Pre-dose (within 60 minutes), 15,30, 45,60,75,90minutes after the beginning of infusion, 15minutes, 30minutes, 1,3,5,8,16,24,36,48,96,168,240,336hours after infusion completed
  Elimination half-life
AUC_%Extrap | Pre-dose (within 60 minutes), 15,30, 45,60,75,90minutes after the beginning of infusion, 15 minutes, 30 minutes, 1,3,5,8,16,24,36,48,96,168,240,336 hours after infusion completed
  Percentage of remaining area，Calculate as [(AUC[0-∞]- AUC[0-t]）/ AUC[0-∞]]×100%
CL/F | Pre-dose (within 60 minutes), 15,30, 45,60,75,90 minutes after the beginning of infusion, 15 minutes, 30 minutes, 1,3,5,8,16,24,36,48,96,168,240,336 hours after infusion completed
  Apparent clearance
Vd/F | Pre-dose (within 60 minutes), 15,30, 45,60,75,90 minutes after the beginning of infusion, 15 minutes, 30 minutes, 1,3,5,8,16,24,36,48,96,168,240,336 hours after infusion completed
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sun Memorial Hospital, Sun Yat-Sun University, Guangzhou, Guangdong, China